CLINICAL TRIAL: NCT07279415
Title: Activate Tennessee: A CHW-Supported Program for Patient Activation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: Baptist Memorial Health Care Corporation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cherokee Health Systems (Unknown)
Responsible Party: Principal Investigator, Stephania T. Miller-Hughes, Professor, Meharry Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TR72217X5599; OT2HL158287 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Hypertension; Cardio Vascular Disease; Infectious Diseases Morbidity; Chronic Kidney Disease; Hypercholesterolemia
Keywords: community health worker, co-morbidities
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Renal Insufficiency, Chronic; Hypercholesterolemia | interventions — Methods; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker Support - Pre-scheduled sessions (Active Comparator)
  Interventions: Behavioral: Intervention
- Community Health Worker Support - Participant-requested sessions (Active Comparator)
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention — Persons assigned to the intervention group will receive strategic and intentional outreach and support from a CHW for 9 months to carry out the patient activation intervention. CHWs will work with persons in the intervention group to develop an Individual Patient Health Activation Plan (IHAP) that is informed by the participants individual health conditions. The IHAP will address priorities and barriers to obtaining optimal health, access to care, and adherence to a health care plan. CHWs will actively outreach the study participant a minimum of monthly to see how they are doing and to update or modify the IHAP, as needed. They will assist the participant in understanding medical advice, developing chronic disease self-management skills, accessing health care, making appointments, and addressing challenges arising from SDoH. CHWs will also utilize motivational interviewing to assist participants in making
  Arms: Community Health Worker Support - Pre-scheduled sessions
Behavioral: Control Group — Persons in the comparator group will receive support to complete an IHAP and access to an interactive community resource website. CHWs will remain available to comparator group participants in response to communicated need and interest but will not provide active outreach to participants.
  Arms: Community Health Worker Support - Participant-requested sessions

SUMMARY:
The research project will involve community health workers (CHWs) that will help participants to better understand their medical conditions and to responsibly manage their medical needs. The project will focus on participants with the greatest medical needs and those that have many different illnesses at the same time. CHWs will help guide participants in focusing on improving their knowledge and confidence to manage their health conditions and to improve their ability to understand how the healthcare system works. This will give participants the opportunity to take charge of their illnesses and possibly improve their health conditions over time. The CHWs will work together with participants to develop a health plan focused on their specific health needs.

DETAILED DESCRIPTION:
Medically underserved persons living with at least two chronic conditions will be recruited for the study.

Participants assigned to the intervention group will receive strategic and intentional outreach and support from a CHW for 9 months to carry out the patient activation intervention. CHWs will work with participants in the intervention group to develop an Individual Patient Health Activation Plan (IHAP) that is informed by the participants individual health conditions and responses to survey questions. CHWs will actively engage in outreach with participants at a minimum of once a month to see how they are doing and to update or modify the IHAP, as needed. They will assist the participant in understanding medical advice, developing chronic disease self-management skills, accessing health care, making appointments, and addressing challenges arising from social determinants of health. CHWs will also utilize motivational interviewing to assist participants in making progress on their activation goals. CHWs will follow up with the study participant monthly but remain available to participants as frequently as participants communicate the need and interest. Beyond the minimum frequency of monthly, the length and frequency of visits will be determined collaboratively based on participant needs and goals. Fidelity will be measured by completion of participant's IHAP and monthly completion of CHW documentation including documented use of at least two patient activation interventions.

Participants in the comparator group will receive support to complete an IHAP and access to an interactive community resource website. CHWs will remain available to comparator group participants in response to communicated need and interest but will not provide active outreach to participants.

Both groups s will meet with the CHWs four times (Baseline, 3 months, 6 months, and 9 months) to complete study surveys and questionnaires, including the patient activation, the primary study outcome.

ELIGIBILITY:
Inclusion criteria:

* 18 years and older,
* Able to speak and understand English
* Have been told by a health care provider that they have two or more, chronic health conditions
* Are classified as medically underserved or socially vulnerable person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure | From enrollment to end of 9 months
  Scored from 0 to 100 with higher scores denoting higher levels of patient activation, it measures participant knowledge, skills, and confidence to manage their own health and healthcare, navigate the healthcare system, and address social barriers that create challenges in their ability to achieve optimal health.

CONTACTS AND LOCATIONS:
Overall Officials: Stephania M Miller-Hughes, PhD, MS, MSCI, Principal Investigator — Meharry Medical College

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 24. Association of State and Territorial Health Officials. (n.d.). Community health workers: evidence of their effectiveness. Association of State and Territorial Health Officials. Accessed on April 10, 2025: https://www.astho.org/globalassets/pdf/community-health-workers-summary-evidence.pdf
- [Background] Kangovi S, Mitra N, Turr L, Huo H, Grande D, Long JA. A randomized controlled trial of a community health worker intervention in a population of patients with multiple chronic diseases: Study design and protocol. Contemp Clin Trials. 2017 Feb;53:115-121. doi: 10.1016/j.cct.2016.12.009. Epub 2016 Dec 10. PMID 27965180
- [Background] Crespo R, Christiansen M, Tieman K, Wittberg R. An Emerging Model for Community Health Worker-Based Chronic Care Management for Patients With High Health Care Costs in Rural Appalachia. Prev Chronic Dis. 2020 Feb 13;17:E13. doi: 10.5888/pcd17.190316. PMID 32053481
- [Background] 21. Patel MI, Kapphahn K, Salava D, et al. The effect of a multilevel community health worker-led intervention on health-related quality of life, patient activation, acute care use, and total costs of care: A randomized controlled trial. Journal of Clinical Oncology. 2022;40(16_suppl):6500-6500.
- [Background] Jana S, Basu I, Rotheram-Borus MJ, Newman PA. The Sonagachi Project: a sustainable community intervention program. AIDS Educ Prev. 2004 Oct;16(5):405-14. doi: 10.1521/aeap.16.5.405.48734. PMID 15491952
- [Background] Liebman AK, Juarez PM, Leyva C, Corona A. A pilot program using promotoras de salud to educate farmworker families about the risk from pesticide exposure. J Agromedicine. 2007;12(2):33-43. doi: 10.1300/J096v12n02_04. PMID 18086652
- [Background] Morgan K, Lee J, Sebar B. Community health workers: a bridge to healthcare for people who inject drugs. Int J Drug Policy. 2015 Apr;26(4):380-7. doi: 10.1016/j.drugpo.2014.11.001. Epub 2014 Nov 13. PMID 25477284
- [Background] Stupplebeen DA, Barnett-Sherrill AT, Sentell TL. Community Health Workers in Hawai'i: A Scoping Review and Framework Analysis of Existing Evidence. Hawaii J Med Public Health. 2019 Jun;78(6 Suppl 1):6-14. PMID 31285962
- [Background] Bellhouse S, McWilliams L, Firth J, Yorke J, French DP. Are community-based health worker interventions an effective approach for early diagnosis of cancer? A systematic review and meta-analysis. Psychooncology. 2018 Apr;27(4):1089-1099. doi: 10.1002/pon.4575. Epub 2017 Nov 23. PMID 29080378
- [Background] Gwede CK, Ashley AA, McGinnis K, Montiel-Ishino FA, Standifer M, Baldwin J, Williams C, Sneed KB, Wathington D, Dash-Pitts L, Green BL. Designing a community-based lay health advisor training curriculum to address cancer health disparities. Health Promot Pract. 2013 May;14(3):415-24. doi: 10.1177/1524839912458675. Epub 2012 Sep 14. PMID 22982709
- [Background] Gilmore B, McAuliffe E. Effectiveness of community health workers delivering preventive interventions for maternal and child health in low- and middle-income countries: a systematic review. BMC Public Health. 2013 Sep 13;13:847. doi: 10.1186/1471-2458-13-847. PMID 24034792
- [Background] Kangovi S, Mitra N, Norton L, Harte R, Zhao X, Carter T, Grande D, Long JA. Effect of Community Health Worker Support on Clinical Outcomes of Low-Income Patients Across Primary Care Facilities: A Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1635-1643. doi: 10.1001/jamainternmed.2018.4630. PMID 30422224
- [Background] Vasan A, Morgan JW, Mitra N, Xu C, Long JA, Asch DA, Kangovi S. Effects of a standardized community health worker intervention on hospitalization among disadvantaged patients with multiple chronic conditions: A pooled analysis of three clinical trials. Health Serv Res. 2020 Oct;55 Suppl 2(Suppl 2):894-901. doi: 10.1111/1475-6773.13321. Epub 2020 Jul 8. PMID 32643163
- [Background] Kim K, Choi JS, Choi E, Nieman CL, Joo JH, Lin FR, Gitlin LN, Han HR. Effects of Community-Based Health Worker Interventions to Improve Chronic Disease Management and Care Among Vulnerable Populations: A Systematic Review. Am J Public Health. 2016 Apr;106(4):e3-e28. doi: 10.2105/AJPH.2015.302987. Epub 2016 Feb 18. PMID 26890177
- [Background] Swider SM. Outcome effectiveness of community health workers: an integrative literature review. Public Health Nurs. 2002 Jan-Feb;19(1):11-20. doi: 10.1046/j.1525-1446.2002.19003.x. PMID 11841678
- [Background] Covert H, Sherman M, Miner K, Lichtveld M. Core Competencies and a Workforce Framework for Community Health Workers: A Model for Advancing the Profession. Am J Public Health. 2019 Feb;109(2):320-327. doi: 10.2105/AJPH.2018.304737. Epub 2018 Dec 20. PMID 30571307
- [Background] Knowles M, Crowley AP, Vasan A, Kangovi S. Community Health Worker Integration with and Effectiveness in Health Care and Public Health in the United States. Annu Rev Public Health. 2023 Apr 3;44:363-381. doi: 10.1146/annurev-publhealth-071521-031648. PMID 37010928
- [Background] Hill-Briggs F, Adler NE, Berkowitz SA, Chin MH, Gary-Webb TL, Navas-Acien A, Thornton PL, Haire-Joshu D. Social Determinants of Health and Diabetes: A Scientific Review. Diabetes Care. 2020 Nov 2;44(1):258-79. doi: 10.2337/dci20-0053. Online ahead of print. No abstract available. PMID 33139407
- [Background] Novilla MLB, Goates MC, Leffler T, Novilla NKB, Wu CY, Dall A, Hansen C. Integrating Social Care into Healthcare: A Review on Applying the Social Determinants of Health in Clinical Settings. Int J Environ Res Public Health. 2023 Oct 2;20(19):6873. doi: 10.3390/ijerph20196873. PMID 37835143
- [Background] Shahid R, Shoker M, Chu LM, Frehlick R, Ward H, Pahwa P. Impact of low health literacy on patients' health outcomes: a multicenter cohort study. BMC Health Serv Res. 2022 Sep 12;22(1):1148. doi: 10.1186/s12913-022-08527-9. PMID 36096793
- [Background] Coughlin SS, Vernon M, Hatzigeorgiou C, George V. Health Literacy, Social Determinants of Health, and Disease Prevention and Control. J Environ Health Sci. 2020;6(1):3061. Epub 2020 Dec 16. No abstract available. PMID 33604453
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] Woolf SH, Braveman P. Where health disparities begin: the role of social and economic determinants--and why current policies may make matters worse. Health Aff (Millwood). 2011 Oct;30(10):1852-9. doi: 10.1377/hlthaff.2011.0685. PMID 21976326
- [Background] Fisher NF, Jampolsky A, Scott AB. Traumatic bitemporal hemianopsia. I. Diagnosis of macular splitting. Am J Ophthalmol. 1968 Feb;65(2):237-42. doi: 10.1016/0002-9394(68)93594-0. No abstract available. PMID 5636025